CLINICAL TRIAL: NCT02704065
Title: Recurrent AA Amyloidosis After Renal Transplantation: Effects on Allograft Survival
Brief Title: Recurrent AA Amyloidosis After Renal Transplantation
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Yasar Caliskan, Associate Professor of Medicine, Istanbul University
Other Study IDs: 32447/199
Record Dates: First submitted 2016-03-04; First posted 2016-03-09 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: AA Amyloidosis
Keywords: amyloidosis; renal transplantation
MeSH Terms: conditions — AA amyloidosis; Amyloidosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Recurrent AA amyloidosis: Renal transplant recipients with biopsy-confirmed AA amyloidosis in the renal allograft
- Control group 1: Renal transplant recipients whose primary diseases are amyloidosis with no clinical or laboratory signs of recurrence in the renal allograft
- Control group 2: Renal transplant recipients whose primary diseases are other than amyloidosis

SUMMARY:
End-stage renal disease related to AA amyloidosis is well characterized but there is limited data concerning patient and graft outcomes after renal transplantation. The aim of this study is to evaluate the clinical features of, and risk factors for recurrent AA amyloidosis, as well as the effects of these factors on the ultimate outcome of renal allografts.

DETAILED DESCRIPTION:
AA amyloidosis is a rare but serious complication of several chronic inflammatory diseases including recurrent hereditary periodic fever syndromes. Although end-stage renal disease related to AA amyloidosis is well characterized, there is limited data concerning patient and graft outcomes after renal transplantation, with most of the findings reported from small series. Recurrence of amyloidosis in the renal allograft might be underdiagnosed, assessing graft and patient outcomes in larger study groups will bring better understanding and new strategies in daily practice.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplantation recipients whose primary renal disease is AA amyloidosis; patients with allograft biopsy-confirmed AA amyloidosis (for study group) and patients with no clinical or laboratory signs of recurrence in the renal allograft (for control group 1)
* Renal transplantation recipients whose primary diseases are other than AA amyloidosis (for control group 2)

Exclusion Criteria:

* Patients who are unwilling or unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Allograft survival | 1 - 5 years

SECONDARY OUTCOMES:
Allograft rejection | 1 - 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yasar Caliskan, MD, Principal Investigator — Division of Nephrology, Department of Internal Medicine, Istanbul Faculty of Medicine
Locations (4):
- Turkey (Türkiye) (4):
  - Division of Nephrology, Department of Internal Medicine, Uludag University Faculty of Medicine, Bursa
  - Division of Nephrology, Department of Internal Medicine, Istanbul Faculty of Medicine, Istanbul
  - Division of Nephrology, Department of Internal Medicine, Cerrahpasa Faculty of Medicine, Istanbul
  - Division of Nephrology, Sisli Hamidiye Etfal Training and Education Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kofman T, Grimbert P, Canoui-Poitrine F, Zuber J, Garrigue V, Mousson C, Frimat L, Kamar N, Couvrat G, Bouvier N, Albano L, Le Thuaut A, Pillebout E, Choukroun G, Couzi L, Peltier J, Mariat C, Delahousse M, Buchler M, Le Pogamp P, Bridoux F, Pouteil-Noble C, Lang P, Audard V. Renal transplantation in patients with AA amyloidosis nephropathy: results from a French multicenter study. Am J Transplant. 2011 Nov;11(11):2423-31. doi: 10.1111/j.1600-6143.2011.03620.x. Epub 2011 Jun 30. PMID 21714848